CLINICAL TRIAL: NCT00421733
Title: VITAL Study - Selective VITamin D Receptor Activator (Paricalcitol) for Albuminuria Lowering Study: A Phase 2, Prospective, Randomized, Double-blind, Placebo-Controlled, Multicenter Study to Evaluate the Safety and Efficacy of Paricalcitol Capsules on Reducing Albuminuria in Type 2 Diabetic Nephropathy Subjects Who Are Currently Being Treated With Renin-angiotensin System Inhibitors
Brief Title: The Effect of Paricalcitol Capsules on Reducing Albuminuria in Patients With Type 2 Diabetic Nephropathy Being Treated With Renin-angiotensin System Inhibitors
Acronym: VITAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M05-741; 2006-001363-31 (EudraCT Number)
Record Dates: First submitted 2007-01-10; First posted 2007-01-12 (Estimated); Results first posted 2010-09-14 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Diabetic Nephropathy; Chronic Kidney Disease
Keywords: Type 2 Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies; Renal Insufficiency, Chronic | interventions — paricalcitol; Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Paricalcitol 1 mcg (Active Comparator): One paricalcitol 1 mcg capsule and one matching placebo capsule per dose
  Interventions: Drug: Zemplar (paricalcitol ) capsules
- Paricalcitol 2 mcg (Active Comparator): Two paricalcitol 1 mcg capsules per dose
  Interventions: Drug: Zemplar (paricalcitol) capsules
- Placebo (Placebo Comparator): Two placebo capsules per dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zemplar (paricalcitol ) capsules — Group 2 - paricalcitol 1 mcg capsules once daily (one paricalcitol 1 mcg capsule once daily and one matching placebo capsule once daily)
  Other Names: ABT-358; paricalcitol; Zemplar
  Arms: Paricalcitol 1 mcg
Drug: Zemplar (paricalcitol) capsules — Group 3 - paricalcitol 2 mcg capsules once daily (two paricalcitol 1 mcg capsules once daily)
  Other Names: ABT-358; paricalcitol; Zemplar
  Arms: Paricalcitol 2 mcg
Drug: Placebo — Group 1 - Placebo once daily (two placebo capsules once daily)
  Arms: Placebo

SUMMARY:
The study objective was to evaluate the safety of paricalcitol capsules and the efficacy of paricalcitol capsules for albuminuria reduction in patients with Chronic Kidney Disease (CKD) who have Type 2 diabetic nephropathy and are receiving optimal angiotensin converting enzyme (ACE) inhibitor and/or angiotensin II receptor blocker (ARB) therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant >= 20 years old.
* Participant has Type 2 Diabetes Mellitus and has been treated with at least one anti-hyperglycemic medication within the 12 months prior to the Screening Phase
* Participant has been receiving a stable dose (i.e., same type and regimen) of ACEi and/or ARB for at least three months prior to the Screening Phase. However, participant may have switched to different brands but at equivalent doses during the three months prior to the Screening Phase.
* Participant is not expected to begin dialysis for at least 6 months.
* If female, participant is not breast feeding or is not pregnant.
* For entry into the Treatment Phase, the participant must satisfy the following criteria based on the Screening laboratory values:

  * Estimated glomerular filtration rate (GFR) between 15-90 mL/min/1.73m2 by simplified Modification in Diet in Renal Disease (MDRD) formula
  * Urinary albumin to creatinine ratio (UACR) between 100 and 3000 mg/g as determined by the mean of the three first morning void urine specimens obtained within one week of each other
  * Corrected serum calcium level <= 9.8 mg/dL
  * intact parathyroid hormone (iPTH) value between 35-500 pg/mL
  * Glycosylated hemoglobin A1c (HbA1c) <= 12%
  * Serum albumin > 3.0 g/dL
  * Negative urine pregnancy test for female participants

Exclusion Criteria:

* Participant has previously been on prescription-based vitamin D therapy within the six months prior to the Screening Phase.
* Participant has a history of an allergic reaction or significant sensitivity to paricalcitol or to drugs similar to the study drug.
* Participant has primary glomerulonephritis or secondary nephritis in addition to diabetic nephropathy.
* Participant has had acute renal failure within 12 weeks of the Screening Phase, defined as an acute rise (of >= 0.5 mg/dL) in serum creatinine to > 4 mg/dL.
* Participant has chronic gastrointestinal disease.
* Participant has secondary hypertension.
* Participant has poorly controlled hypertension.
* Participant has a history of kidney stones.
* Participant has a history of drug or alcohol abuse within six months prior to the Screening Phase.
* Participant has evidence of poor compliance with diet or medication.
* Participant has received any investigational drug within 30 days prior to study drug administration.
* Participant is taking calcitonin, bisphosphonates, cinacalcet, glucocorticoids (except topical glucocorticoids), or other drugs that may affect calcium, or bone metabolism, other than calcium containing phosphate binder or female participants on stable (same dose and product for three months) estrogen and/or progestin therapy.
* For any reason, participant is considered by the Investigator to be an unsuitable candidate to receive paricalcitol capsules or is put at risk by study procedures.
* Participant is known to be human immunodeficiency virus (HIV) positive.
* Participant has used known inhibitors or inducers of cytochrome P450 3A (CYP3A) within two weeks prior to study drug administration.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2006-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Andress, MD, Study Director — Abbott
Locations (72):
- United States (27):
  - Site Reference ID/Investigator# 862, Phoenix, Arizona
  - Site Reference ID/Investigator# 864, Fountain Valley, California
  - Site Reference ID/Investigator# 7291, Yuba City, California
  - Site Reference ID/Investigator# 853, Hudson, Florida
  - Site Reference ID/Investigator# 867, Lauderdale Lakes, Florida
  - Site Reference ID/Investigator# 857, Pembroke Pines, Florida
  - Site Reference ID/Investigator# 8901, West Palm Beach, Florida
  - Site Reference ID/Investigator# 7113, Roswell, Georgia
  - Site Reference ID/Investigator# 2531, Chicago, Illinois
  - Site Reference ID/Investigator# 3371, Evanston, Illinois
  - Site Reference ID/Investigator# 869, Indianapolis, Indiana
  - Site Reference ID/Investigator# 8054, Baton Rouge, Louisiana
  - Site Reference ID/Investigator# 854, Rockville, Maryland
  - Site Reference ID/Investigator# 6281, Boston, Massachusetts
  - Site Reference ID/Investigator# 859, Brooklyn Center, Minnesota
  - Site Reference ID/Investigator# 7214, Omaha, Nebraska
  - Site Reference ID/Investigator# 8046, Albany, New York
  - Site Reference ID/Investigator# 866, Charlotte, North Carolina
  - Site Reference ID/Investigator# 8039, Greenville, North Carolina
  - Site Reference ID/Investigator# 8053, Morehead City, North Carolina
  - Site Reference ID/Investigator# 6626, Winston-Salem, North Carolina
  - Site Reference ID/Investigator# 7495, Carlisle, Pennsylvania
  - Site Reference ID/Investigator# 9061, Dallas, Texas
  - Site Reference ID/Investigator# 8325, Dallas, Texas
  - Site Reference ID/Investigator# 856, Dallas, Texas
  - Site Reference ID/Investigator# 7494, San Antonio, Texas
  - Site Reference ID/Investigator# 774, San Antonio, Texas
- Germany (3):
  - Site Reference ID/Investigator# 6316, Düsseldorf
  - Site Reference ID/Investigator# 5167, Hanover
  - Site Reference ID/Investigator# 6302, Ludwigshafen
- Greece (4):
  - Site Reference ID/Investigator# 6314, Athens
  - Site Reference ID/Investigator# 6306, Ioannina
  - Site Reference ID/Investigator# 5631, Thessaloniki
  - Site Reference ID/Investigator# 6310, Thessaloniki
- Italy (4):
  - Site Reference ID/Investigator# 6312, Bergamo
  - Site Reference ID/Investigator# 6303, Brescia
  - Site Reference ID/Investigator# 6309, Milan
  - Site Reference ID/Investigator# 6210, Modena
- Site Reference ID/Investigator# 6207, Groningen, Netherlands
- Poland (4):
  - Site Reference ID/Investigator# 6304, Bydgoszcz
  - Site Reference ID/Investigator# 5622, Katowice
  - Site Reference ID/Investigator# 5203, Szczecin
  - Site Reference ID/Investigator# 6315, Warsaw
- Portugal (2):
  - Site Reference ID/Investigator# 6327, Lisbon
  - Site Reference ID/Investigator# 6326, Porto
- Puerto Rico (15):
  - Site Reference ID/Investigator# 6916, Caguas
  - Site Reference ID/Investigator# 5175, Carolina
  - Site Reference ID/Investigator# 6290, Las Piedras
  - Site Reference ID/Investigator# 5179, Ponce
  - Site Reference ID/Investigator# 6293, Ponce
  - Site Reference ID/Investigator# 5173, Ponce
  - Site Reference ID/Investigator# 6300, Ponce
  - Site Reference ID/Investigator# 5168, Ponce
  - Site Reference ID/Investigator# 7298, Rio Piedras
  - Site Reference ID/Investigator# 5170, San Juan
  - Site Reference ID/Investigator# 7509, San Juan
  - Site Reference ID/Investigator# 6288, San Juan
  - Site Reference ID/Investigator# 6291, San Juan
  - Site Reference ID/Investigator# 6919, Toa Baja
  - Site Reference ID/Investigator# 6296, Yabucoa
- Spain (7):
  - Site Reference ID/Investigator# 6569, Barcelona
  - Site Reference ID/Investigator# 10621, Galdakao
  - Site Reference ID/Investigator# 6330, L'Hospitalet de
  - Site Reference ID/Investigator# 5111, Madrid
  - Site Reference ID/Investigator# 5110, Oviedo
  - Site Reference ID/Investigator# 6329, Santander
  - Site Reference ID/Investigator# 11281, Valencia
- Taiwan (5):
  - Site Reference ID/Investigator# 8335, Taichung
  - Site Reference ID/Investigator# 7927, Taichung
  - Site Reference ID/Investigator# 6294, Taipei
  - Site Reference ID/Investigator# 6285, Taipei
  - Site Reference ID/Investigator# 6286, Xinzhuang

REFERENCES:
- [Derived] Coyne DW, Andress DL, Amdahl MJ, Ritz E, de Zeeuw D. Effects of paricalcitol on calcium and phosphate metabolism and markers of bone health in patients with diabetic nephropathy: results of the VITAL study. Nephrol Dial Transplant. 2013 Sep;28(9):2260-8. doi: 10.1093/ndt/gft227. Epub 2013 Jun 19. PMID 23787544
- [Derived] de Zeeuw D, Agarwal R, Amdahl M, Audhya P, Coyne D, Garimella T, Parving HH, Pritchett Y, Remuzzi G, Ritz E, Andress D. Selective vitamin D receptor activation with paricalcitol for reduction of albuminuria in patients with type 2 diabetes (VITAL study): a randomised controlled trial. Lancet. 2010 Nov 6;376(9752):1543-51. doi: 10.1016/S0140-6736(10)61032-X. PMID 21055801

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paricalcitol 1 Mcg | Paricalcitol 2 Mcg | Placebo
Started | 93 | 95 | 93
Completed | 78 | 69 | 73
Not Completed | 15 | 26 | 20
Not completed — Adverse Event | 4 | 9 | 2
Not completed — Lost to Follow-up | 1 | 2 | 4
Not completed — Withdrawal by Subject | 1 | 2 | 7
Not completed — Death | 0 | 3 | 0
Not completed — Required dialysis | 1 | 0 | 0
Not completed — Administrative | 2 | 0 | 0
Not completed — Did not satisfy entry criteria | 1 | 3 | 2
Not completed — Sponsor request | 1 | 0 | 3
Not completed — Protocol deviation | 4 | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paricalcitol 1 Mcg | Paricalcitol 2 Mcg | Placebo | Total
Number analyzed (Participants) | 93 | 95 | 93 | 281
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 45 | 47 | 44 | 136
  >=65 years | 48 | 48 | 49 | 145
Age Continuous [Mean (Standard Deviation); unit: years] | 64.0 (10.15) | 64.7 (9.92) | 64.5 (11.23) | 64.4 (10.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 26 | 33 | 86
  Male | 66 | 69 | 60 | 195
Region of Enrollment [Number; unit: participants]
  Portugal | 2 | 2 | 0 | 4
  United States | 57 | 60 | 64 | 181
  Taiwan | 10 | 14 | 10 | 34
  Greece | 1 | 3 | 1 | 5
  Poland | 4 | 4 | 4 | 12
  Spain | 11 | 3 | 9 | 23
  Netherlands | 0 | 0 | 1 | 1
  Germany | 4 | 8 | 1 | 13
  Italy | 4 | 1 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to the Last On-treatment Measurement in Urine Albumin to Creatinine Ratio (UACR) Levels Determined From the First Morning Void (FMV) Urine Collections Comparing Placebo to the Combined Paricalcitol Treatment Groups (1 Mcg and 2 Mcg).
Description: UACR is defined as the ratio: milligram of albumin per gram of creatinine. Baseline UACR was determined as the mean of the 3 UACR measurements from FMV urine collections obtained within 1 week prior to the day of the first dose of study drug. The last on-treatment measurement was the mean of the 3 UACR measurements obtained from FMV urine collections obtained within 1 week of the final week of treatment. The UACR data were log transformed prior to analysis.
Time Frame: Baseline (within 1 week prior to first treatment) through 24 weeks of treatment
Population: Intent-to-treat population, which was all randomized participants who received at least 1 dose of study drug. Subjects without both a baseline and last on-treatment measurement were excluded from the primary efficacy analysis. As such, sample size was N=88 for placebo, N=92 for 1 mcg and for 2 mcg paricalcitol, and N=184 for combined paricalcitol.
Measure: Mean (Standard Deviation); unit: log milligram/gram creatinine
Groups:
- Placebo: Two placebo capsules per dose (N=88)
- Combined Paricalcitol 1 Mcg and 2 Mcg: Combined participants in the 1 mcg and 2 mcg paricalcitol groups (N=92+92=184).
Arm/Group | Placebo | Combined Paricalcitol 1 Mcg and 2 Mcg | Paricalcitol 1 Mcg | Paricalcitol 2 Mcg
Number analyzed (Participants) | 88 | 184 | 92 | 92
log milligram/gram creatinine | -0.03 (0.61) | -0.18 (0.70) | -0.15 (0.72) | -0.22 (0.69)
Statistical Analysis 1: Comparison: Placebo vs Combined Paricalcitol 1 Mcg and 2 Mcg; Test type: Superiority or Other; p = 0.071, ANCOVA — There were no P-value adjustments for multiple comparisons; 1-way ANCOVA using treatment group as the factor and baseline FMV UACR as the covariate
Statistical Analysis 2: Comparison: Placebo vs Paricalcitol 1 Mcg; Test type: Superiority or Other; p = 0.229, ANCOVA — There were no P-value adjustments for multiple comparisons; 1-way ANCOVA with treatment group as the factor and baseline FMV UACR as the covariate
Statistical Analysis 3: Comparison: Placebo vs Paricalcitol 2 Mcg; Test type: Superiority or Other; p = 0.053, ANCOVA — There were no P-value adjustments for multiple comparisons; 1-way ANCOVA using treatment group as the factor and baseline FMV UACR as the covariate

2. Secondary Outcome: Number of Participants Achieving a 15% or Greater Reduction From Baseline to Last On-treatment Urine Albumin to Creatinine Ratio (UACR) Levels.
Description: Number of participants whose last on-treatment albumin to creatinine ratio (UACR) value was reduced at least 15% from the baseline value. Albumin values were determined from 24-hour urine collections from the baseline and last on-treatment visits.
Time Frame: Baseline (within 1 week prior to first treatment) through 24 weeks of treatment
Population: Intent-to-treat population, which was all randomized subjects who received at least one dose of study drug. Subjects who did not have both a baseline measurement and a last on-treatment visit value were excluded from the analyses.
Measure: Number; unit: Participants
Arm/Group | Paricalcitol 1 Mcg | Paricalcitol 2 Mcg | Placebo
Number analyzed (Participants) | 92 | 92 | 88
Participants | 48 | 51 | 35
Statistical Analysis 1: Comparison: Paricalcitol 1 Mcg vs Placebo; Test type: Superiority or Other; p = 0.102, Fisher Exact
Statistical Analysis 2: Comparison: Paricalcitol 2 Mcg vs Placebo; Test type: Superiority or Other; p = 0.038, Fisher Exact

3. Secondary Outcome: Change From Baseline to the Last On-treatment Measurement in Albumin Levels Determined From 24-hour Urine Collection.
Description: The change is mean change from baseline to the last on-treatment value, with the data being log transformed prior to analysis. Albumin values were determined from 24-hour urine collections from the baseline and last on-treatment visits.
Time Frame: Baseline (within 1 week prior to first treatment) through 24 weeks of treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: log milligrams of albumin per 24 hours
Arm/Group | Paricalcitol 1 Mcg | Paricalcitol 2 Mcg | Placebo
Number analyzed (Participants) | 74 | 72 | 78
log milligrams of albumin per 24 hours | -0.10 (0.73) | -0.44 (0.90) | -0.08 (0.73)
Statistical Analysis 1: Comparison: Paricalcitol 1 Mcg vs Placebo; Test type: Superiority or Other; p = 0.855, ANCOVA; 2-way ANCOVA: baseline UACR as covariate; fixed factors for treatment group, stratification level, and treatment by stratification level interaction; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.26 to 0.22]
Statistical Analysis 2: Comparison: Paricalcitol 2 Mcg vs Placebo; Test type: Superiority or Other; p = 0.009, ANCOVA; [statistical method as in outcome 3, analysis 1]; Mean Difference (Net) = -0.33, 95% CI 2-sided [-0.57 to -0.08]

4. Secondary Outcome: Change From Baseline to the Last On-treatment Observation in Intact Parathyroid Hormone (iPTH) Levels.
Description: Change is mean change in picograms of iPTH per milliliter of serum.
Time Frame: Baseline (screening period) through 24 weeks of treatment
Population: Intent-to-treat population, which was all randomized subjects who received at least one dose of study drug. Subjects who did not have both a baseline and a last on-treatment measurement were excluded from the analyses.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Paricalcitol 1 Mcg | Paricalcitol 2 Mcg | Placebo
Number analyzed (Participants) | 92 | 90 | 88
picogram/milliliter | -26.7 (55.2) | -50.7 (63.1) | 18.3 (55.3)
Statistical Analysis 1: Comparison: Paricalcitol 1 Mcg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; 1-way ANCOVA with treatment group as the factor and baseline iPTH as covariate
Statistical Analysis 2: Comparison: Paricalcitol 2 Mcg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; 1-way ANCOVA with treatment group as the factor and baseline iPTH as covariate

ADVERSE EVENTS:
Time Frame: up to 24 weeks
Description: Treatment-emergent serious adverse and non-serious adverse events were reported after the first dose of study drug through 30 days after the last dose of study drug.
Arm/Group | Paricalcitol 1 Mcg | Paricalcitol 2 Mcg | Placebo
Serious Adverse Events (participants affected / at risk) | 13/93 | 19/95 | 12/93
Other Adverse Events (participants affected / at risk) | 38/93 | 46/95 | 46/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol 1 Mcg (N=93) | Paricalcitol 2 Mcg (N=95) | Placebo (N=93)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Gastrointestinal angiodysplasia haemorrhagic (Congenital, familial and genetic disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Retinal oedema (Eye disorders) | 1 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Asthenia (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0
Death (General disorders) | 0 | 1 | 0
Impaired healing (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 0
Posteroperative wound infection (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Benign colonic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Oesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 1 | 0
Substance abuse (Psychiatric disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 2 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 1 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Extremity necrosis (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 2 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol 1 Mcg (N=93) | Paricalcitol 2 Mcg (N=95) | Placebo (N=93)
Anemia (Blood and lymphatic system disorders) | 5 | 8 | 5
Constipation (Gastrointestinal disorders) | 3 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 6
Nausea (Gastrointestinal disorders) | 2 | 2 | 4
Chest pain (General disorders) | 0 | 0 | 3
Fatigue (General disorders) | 1 | 5 | 1
Oedema (General disorders) | 3 | 3 | 1
Oedema peripheral (General disorders) | 5 | 4 | 4
Pyrexia (General disorders) | 0 | 0 | 3
Bronchitis (Infections and infestations) | 3 | 2 | 1
Nasopharyngitis (Infections and infestations) | 2 | 3 | 2
Tinea pedis (Infections and infestations) | 0 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 5 | 5 | 4
Urinary tract infection (Infections and infestations) | 2 | 6 | 2
Blood parathyroid hormone decreased (Investigations) | 2 | 3 | 0
Gout (Metabolism and nutrition disorders) | 1 | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 5 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2 | 3
Dizziness (Nervous system disorders) | 3 | 3 | 1
Headache (Nervous system disorders) | 0 | 3 | 4
Chronic obstructive pulmonsry disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 3
Hypertension (Vascular disorders) | 5 | 8 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.